CLINICAL TRIAL: NCT03859063
Title: A Multimodal Individualized Intervention to Prevent Functional Decline After Stroke. A Randomized Controlled Trial on Long-term Follow-up After Stroke (The LAST-long Trial)
Brief Title: Long-term Follow-up After Stroke (The LAST-long Trial)
Acronym: LAST-long
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital, Akershus (Other); Asker & Baerum Hospital (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018/1809
Record Dates: First submitted 2019-02-11; First posted 2019-03-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Rehabilitation; Cognition; Physical Fitness; Case Managers; Secondary prevention
MeSH Terms: conditions — Stroke | interventions — Methods

STUDY DESIGN:
Intervention Model Description: A two armed parallel group randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-blinded. The investigator and outcomes assessor will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Regular follow up by a community based stroke coordinator
  Interventions: Behavioral: Intervention
- Control (Active Comparator): Usual care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — Participants randomized to the intervention arm will be followed with monthly meetings by a stroke coordinator for 18 months. The stroke coordinator will assess the patients risk factors within the domains of physical function, cognitive function, social function, medication and lifestyle factors and make a treatment plan targeting the individual needs for further follow-up.
  Arms: Intervention
Behavioral: Control — Community based follow-up as usual
  Other Names: Usual care
  Arms: Control

SUMMARY:
Despite the improved treatment of acute stroke over the past decades, those suffering from stroke still are at an increased risk of functional and cognitive decline in the long term. The most common consequences of stroke are functional impairments, cognitive impairments, depression and fatigue. These are also regarded as barriers to achieve optimal adherence to the guidelines regarding secondary prevention. The primary aim of this project is to evaluate the effectiveness of a multimodal individualized intervention to prevent functional decline in the long term after stroke.

DETAILED DESCRIPTION:
In a clinical randomized controlled trial, participants randomized to the intervention arm will be followed with monthly meetings by a stroke coordinator for 18 months.

The stroke coordinator will assess the patients risk factors within the domains of physical function, cognitive function, social function, medication and lifestyle factors and make a treatment plan targeting the individual needs for further follow-up.

Those randomized to the control group will receive standard care.

Patients living in the municipalities of Trondheim, Lørenskog and Skedsmo admitted to Akershus University Hospital or St. Olavs University Hospital will be included at the outpatients clinic 3 months after the stroke.

All patients will be re-assessed at 6, 12 and 18 months after inclusion. Primary outcome will be modified Rankin Scale at 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of first ever or recurrent stroke (ischemic stroke or hemorrhage)
* mRS < 5
* Living in Trondheim, Skedsmo or Lørenskog municipality
* Less than 10 points on Short Physical Performance Battery (SPPB) OR less than 26 points on Montreal Cognitive Assessment (MoCA) OR more than 27 points on the 7 item version of the Fatigue Severity Scale (FSS-7) OR more than 7 points on the depression or anxiety items on Hospital Anxiety and Depression Scale (HADS) OR reduced hand function (i.e. fails on Motor Assessment Scale - Advanced arm- and hand function, item 3)
* Able to understand Norwegian
* Able and willing to sign informed consent.

Exclusion Criteria:

* Life expectancy < 12 months
* Other serious diseases, judged by the medical doctor to make it difficult to comply with the intervention (i.e. serious neurological diseases or drug abuse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 18 months
  mRS is an ordinal scale ranging from 0 to 6 measuring global function. 0 denotes no symptoms while 6 denotes death.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | 6 months
  mRS is an ordinal scale ranging from 0 to 6 measuring global function. 0 denotes no symptoms while 6 denotes death.
Modified Rankin Scale (mRS) | 12 months
  mRS is an ordinal scale ranging from 0 to 6 measuring global function. 0 denotes no symptoms while 6 denotes death.
Barthel Index | 6 months
  ADL function
Barthel Index | 12 months
  ADL function
Barthel Index | 18 months
  ADL function
Nottingham IADL | 6 months
  Extended activities of daily life (ADL) function
Nottingham IADL | 12 months
  Extended activities of daily life (ADL) function
Nottingham IADL | 18 months
  Extended activities of daily life (ADL) function
Stroke Impact Scale (SIS) | 6 months
  SIS is a stroke specific quality of life measure, that measures self perceived health within nine domains. The scale within each domain range from 0 to 100 and higher score denotes better health.
Stroke Impact Scale (SIS) | 12 months
  SIS is a stroke specific quality of life measure, that measures self perceived health within nine domains. The scale within each domain range from 0 to 100 and higher score denotes better health.
Stroke Impact Scale (SIS) | 18 months
  SIS is a stroke specific quality of life measure, that measures self perceived health within nine domains. The scale within each domain range from 0 to 100 and higher score denotes better health.
The 5-level EQ-5D version (EQ-5D-5L) | 6 months
  EQ-5D-5L is a generic quality of life measure reporting self perceived health within five domains.
The 5-level EQ-5D version (EQ-5D-5L) | 12 months
  EQ-5D-5L is a generic quality of life measure reporting self perceived health within five domains.
The 5-level EQ-5D version (EQ-5D-5L) | 18 months
  EQ-5D-5L is a generic quality of life measure reporting self perceived health within five domains.
Short Physical Performance Battery (SPPB) | 6 months
  SPPB is a composite scale measuring gait and balance. The scale ranges from 0 to 12 points. Higher score denotes better function.
Short Physical Performance Battery (SPPB) | 12 months
  SPPB is a composite scale measuring gait and balance. The scale ranges from 0 to 12 points. Higher score denotes better function.
Short Physical Performance Battery | 18 months
  SPPB is a composite scale measuring gait and balance. The scale ranges from 0 to 12 points. Higher score denotes better function.
Dynamometer | 6 months
  Grip strength
Dynamometer | 12 months
  Grip strength
Dynamometer | 18 months
  Grip strength
6 Minute Walk Test | 6 months
  Endurance. Walking distance during 6 minutes.
6 Minute Walk Test | 12 months
  Endurance. Walking distance during 6 minutes.
6 Minute Walk Test | 18 months
  Endurance. Walking distance during 6 minutes.
ActivPAL | 6 months
  Activity monitoring across seven days
ActivPAL | 12 months
  Activity monitoring across seven days
ActivPAL | 18 months
  Activity monitoring across seven days
Montreal Cognitive Assessment | 6 months
  Cognitive function
Montreal Cognitive Assessment | 12 months
  Cognitive function
Montreal Cognitive Assessment | 18 months
  Cognitive function
Trail making test A and B | 6 months
  Executive function
Trail making test A and B | 12 months
  Executive function
Trail making test A and B | 18 months
  Executive function
Global Deterioration Scale (GDS) | 6 months
  GDS is a measure of global cognitive function. A score of 1 denotes no symptoms while a score of 7 denotes serious dementia.
Global Deterioration Scale (GDS) | 12 months
  GDS is a measure of global cognitive function. A score of 1 denotes no symptoms while a score of 7 denotes serious dementia.
Global Deterioration Scale (GDS) | 18 months
  GDS is a measure of global cognitive function. A score of 1 denotes no symptoms while a score of 7 denotes serious dementia.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Hospital Anxiety and Depression Scale (HADS) | 12 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Hospital Anxiety and Depression Scale (HADS) | 18 months
  The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Fatigue Severity Scale (FSS-7) | 6 months
  The seven item version of Fatigue Severity Scale is a method of evaluating the impact of fatigue. FSS-7 contains seven statements that rate the severity of fatigue. Each item is scored from 1 to 7. Higher score is indicating more fatigue.
Fatigue Severity Scale (FSS-7) | 12 months
  The seven item version of Fatigue Severity Scale is a method of evaluating the impact of fatigue. FSS-7 contains seven statements that rate the severity of fatigue. Each item is scored from 1 to 7. Higher score is indicating more fatigue.
Fatigue Severity Scale (FSS-7) | 18 months
  The seven item version of Fatigue Severity Scale is a method of evaluating the impact of fatigue. FSS-7 contains seven statements that rate the severity of fatigue. Each item is scored from 1 to 7. Higher score is indicating more fatigue.
Part 2 of the Client Service Receipt Inventory | 6 months
  A measure of caregivers work participation and absenteeism
Part 2 of the Client Service Receipt Inventory | 12 months
  A measure of caregivers work participation and absenteeism
Part 2 of the Client Service Receipt Inventory | 18 months
  A measure of caregivers work participation and absenteeism
Total cholesterol | 6 months
  The level of total cholesterol will be measured by a blood test
Total cholesterol | 12 months
  The level of total cholesterol will be measured by a blood test
Total cholesterol | 18 months
  The level of total cholesterol will be measured by a blood test
Low Density Lipoprotein (LDL) | 6 months
  The LDL level will be measured by a blood test
Low Density Lipoprotein (LDL) | 12 months
  The LDL level will be measured by a blood test
Low Density Lipoprotein (LDL) | 18 months
  The LDL level will be measured by a blood test
High Density Lipoprotein (HDL) | 6 months
  The HDL level will be measured by a blood test
High Density Lipoprotein (HDL) | 12 months
  The HDL level will be measured by a blood test
High Density Lipoprotein (HDL) | 18 months
  The HDL level will be measured by a blood test
Longterm blood sugar (HbA1c) | 6 months
  The HbA1c level will be measured by a blood test
Longterm blood sugar (HbA1c) | 12 months
  The HbA1c level will be measured by a blood test
Longterm blood sugar (HbA1c) | 18 months
  The HbA1c level will be measured by a blood test
Hemoglobin | 6 months
  The hemoglobin level will be measured by a blood test
Hemoglobin | 12 months
  The hemoglobin level will be measured by a blood test
Hemoglobin | 18 months
  The hemoglobin level will be measured by a blood test
Creatinine | 6 months
  The creatinine level will be measured by a blood test
Creatinine | 12 months
  The creatinine level will be measured by a blood test
Creatinine | 18 months
  The creatinine level will be measured by a blood test
C-reactive protein (CRP) | 6 months
  The CRP level will be measured by a blood test
C-reactive protein (CRP) | 12 months
  The CRP level will be measured by a blood test
C-reactive protein (CRP) | 18 months
  The CRP level will be measured by a blood test
Blood pressure | 6 months
  Systolic and diastolic blood pressure will be measured by use of a sphygmomanometer
Blood pressure | 12 months
  Systolic and diastolic blood pressure will be measured by use of a sphygmomanometer
Blood pressure | 18 months
  Systolic and diastolic blood pressure will be measured by use of a sphygmomanometer
Body mass index (BMI) | 6 months
  BMI calculated as kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared
Body mass index (BMI) | 12 months
  BMI calculated as kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared
Body mass index (BMI) | 18 months
  BMI calculated as kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared
Health care costs | 18 months
  Data from available registries will be used to estimate costs in Euro
Adherence to the intervention | 18 months
  Number of attended meetings with the stroke coordinator
Exercise Adherence Rating Scale | 18 months
  Exercise Adherence Rating Scale measures the level of adherence to the recommended and agreed activities and the reasons for not adhering.
Patient diaries | 18 months
  Adherence to the recommended and agreed activities
Adverse events | 18 months
  Adverse events will be registered to assess the safety of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Helbostad, phd prof, Study Director — Norwegian University for Science and Technology
Locations (4):
- Norway (4):
  - Ålesund Hospital, Ålesund
  - Akershus University Hospital, Lørenskog
  - Vestre Viken Bærum Hospital, Sandvika
  - St Olavs Hospital Stroke Unit, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Askim T, Langlo SR, Bergh E, Dohl O, Ellekjaer H, Hokstad A, Ihle-Hansen H, Indredavik B, Lydersen S, Luzum G, Seljeseth Y, Skandsen T, Saltvedt I, Thommessen B. A multimodal individualized long-term intervention to prevent functional decline after stroke (LAST-long): a single blinded randomised controlled trial. Lancet Reg Health Eur. 2025 Nov 13;61:101531. doi: 10.1016/j.lanepe.2025.101531. eCollection 2026 Feb. PMID 41323876
- [Derived] Askim T, Hokstad A, Bergh E, Dohl O, Ellekjaer H, Ihle-Hansen H, Indredavik B, Leer ASM, Lydersen S, Saltvedt I, Seljeseth Y, Thommessen B. Multimodal individualised intervention to prevent functional decline after stroke: protocol of a randomised controlled trial on long-term follow-up after stroke (LAST-long). BMJ Open. 2023 May 10;13(5):e069656. doi: 10.1136/bmjopen-2022-069656. PMID 37164457
- [Derived] Gibson E, Koh CL, Eames S, Bennett S, Scott AM, Hoffmann TC. Occupational therapy for cognitive impairment in stroke patients. Cochrane Database Syst Rev. 2022 Mar 29;3(3):CD006430. doi: 10.1002/14651858.CD006430.pub3. PMID 35349186